CLINICAL TRIAL: NCT01638117
Title: Phase I Clinical Trial to Investigate the Cumulative Skin Irritation of PAC-14028 in Healthy Volunteers
Brief Title: Cumulative Irritation Test of PAC-14028 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AP-TRPV1_PI-02
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium Chloride; Gene Expression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PAC14028-Vehicle (Placebo Comparator): PAC-14028 Cream Vehicle
  Interventions: Other: PAC14028-Vehicle
- PAC14028-0.1 (Experimental): PAC-14028 Cream 0.1%
  Interventions: Drug: PAC14028-0.1
- PAC14028-0.3 (Experimental): PAC-14028 Cream 0.3%
  Interventions: Drug: PAC14028-0.3
- PAC14028-1.0 (Experimental): PAC-14028 Cream 1%
  Interventions: Drug: PAC14028-1.0
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Saline
- Positive control (Active Comparator): Sodium Lauryl Sulfate, 0.5%
  Interventions: Other: Positive

INTERVENTIONS:
Other: PAC14028-Vehicle — PAC-14028 Cream Vehicle, Daily for up to 21 days
  Other Names: PAC-14208 cream vehicle
  Arms: PAC14028-Vehicle
Drug: PAC14028-0.1 — PAC-14028 Cream, 0.1%, Daily for up to 21 days
  Other Names: PAC-14208 Cream 0.1%
  Arms: PAC14028-0.1
Drug: PAC14028-0.3 — PAC-14028 Cream, 0.3%, Daily for up to 21 days
  Other Names: PAC-14208 Cream 0.3%
  Arms: PAC14028-0.3
Drug: PAC14028-1.0 — PAC-14028 Cream, 1%, Daily for up to 21 days
  Other Names: PAC-14028 Cream 1.0%
  Arms: PAC14028-1.0
Other: Saline — Saline, Daily for up to 21 days
  Other Names: 0.9% Sodium chloride
  Arms: Placebo
Other: Positive — Sodium Lauryl Sulfate, 0.5%, Daily for up to 21 days
  Arms: Positive control

SUMMARY:
The purpose of this study is to determine the cumulative irritation potential of the products listed by the Sponsor.

DETAILED DESCRIPTION:
Healthy, adult volunteers of either sex will be patched daily on his/her arm with multiple strengths of PAC-14028 cream, non-active comparator and an active comparator over the course of 21 consecutive days. Twenty-four hours after each application, the Finn-chamber patches will be removed and the site evaluated using a five-point scale for irritation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of either sex, at least 20 years to 59 Years.
* Females must be of non-childbearing potential (i.e., post-menopausal or surgically sterile). All females must submit to a urine pregnancy test and have a negative result at Day 1 and at the final study visit.
* Subjects may be of any skin type or race providing their degree of skin pigmentation does not interfere with readings of skin reactions.
* Who voluntarily decides study participation after receiving detailed explanation about the study and fully understanding it and who provides written consent for compliance with study requirement including proper contraception.

Exclusion Criteria:

* Atopic dermatitis/eczema, psoriasis will be excluded. Any skin disease that would in any way confound interpretation of the study results.
* Asthma and chronic bronchitis will be excluded.
* Inability to evaluate the skin in and around the potential patch test sites on the arm due to erythema, eschar, excoriation, tattoos, scars, unevenness in skin tones, or other skin damage or abnormality.
* A history of sensitivity to any component of any of the formulations and the Finn chamber.
* Used systemic or topical corticosteroids or other immunosuppressive medications within 1 weeks of the Day 1 visit.
* Used nonsteroidal anti-inflammatory medications within 2 weeks of the Day 1 visit.
* Received immunizations within 2 weeks of the Day 1 visit.
* Any major illness within 4 weeks of the Day 1 visit.
* Female who is pregnant, trying to become pregnant, or breast feeding
* Use of chronic medications (such as antihistamines, corticosteroids, analgesics and anti-inflammatories) for one week before and during the study.
* Currently using any medication that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Irritation Score (5-point scale, 0-4) | Daily for 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Han Kim, M.D.,Ph.D., Study Director — Seoul National University Hospital, Department of Dermatology
Locations (1):
- Seoul National University Hospital, Department of Dermatology, Seoul, Seoul, South Korea